CLINICAL TRIAL: NCT04469868
Title: Prospective Study of No Opioids PrescrIptions On Discharge After Surgery (NOPIOiDS)
Brief Title: No Opioids PrescrIptions On Discharge After Surgery
Acronym: NOPIOiDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Badar M. Mian, Professor of Surgery, Albany Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5866
Record Dates: First submitted 2020-07-08; First posted 2020-07-14 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Opioid Use; Prescription Drug Abuse and Dependency; Surgery; Postoperative Pain
Keywords: Opioids; Prescriptions; Surgery; Recovery; Pain score
MeSH Terms: conditions — Substance-Related Disorders; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: All patients who undergo major urologic oncology surgery will be eligible to be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No opioids prescriptions at discharge (Experimental): Patients will receive non-opioid analgesia, mostly over the counter, medications such as acetaminophen or ibuprofen. Opioids may be prescribed if the patients experience break through pain and call the office.
  Interventions: Behavioral: No opioids at discharge

INTERVENTIONS:
Behavioral: No opioids at discharge — Patients who are being scheduled for any major urologic cancer surgery (open or laparoscopic) will be counselled regarding post-operative pain and measures taken during surgery and during hospital stay.
  They will be provided written information on these pain mitigation efforts and the adverse effects associated with opioids use and outpatient prescriptions.
  Patients will be discharged from the hospital without any opioids prescriptions and instructions to use non-opioids analgesics.
  Patients will complete a visual analog pain scale daily for 7 days after discharge from the hospital.
  Patients will be able to call the clinic at anytime for any post-operative pain issues.

SUMMARY:
Opioid analgesics are routinely prescribed for these patients for post-operative pain control. Even a short exposure to opioids in opioid-naïve patients following minor or major surgery has been associated with de novo habitual or persistent use of opioids in 5-30% of patients. The goal of the study to eliminate the use of outpatient opioids prescriptions after major urologic surgery.

DETAILED DESCRIPTION:
Nearly 200 million opioid prescriptions are dispensed per year in the United States. Opioid prescriptions given by medical providers are a major contributor to the opioid abuse epidemic. Nearly 40% of opioid overdose-related deaths occur due to prescribed opioids. Among patients diagnosed with opiate dependence, 80% had received an opioid prescription prior to their abuse diagnosis and 51% had a family member who had an opioid prescription, Thus, opioids prescriptions, which are often in excess of the need by the patient, are a major contributor to this public health crisis.

The investigators devised a prospective intervention study to eliminate or significantly reduced the use of opioids prescribed at hospital discharge after major urologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing major urologic cancer surgery, either open or laparoscopic, will be included in the study.
* This will include all open or laparoscopic or robotic surgery including radical prostatectomy, radical cystectomy, radical nephrectomy, partial nephrectomy, nephron-ureterectomy, and similar procedures.

Exclusion Criteria:

* Those with allergy or intolerance to NSAIDS may be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Opioids prescribing at hospital discharge | 30 days
  Patients will be discharged with no or few opioids after surgery along with instruction on how to use non-opioid analgesic measures.
All opioids prescriptions within 30 days of surgery | 30 days
  The electronic medical records and pharmacy records will be monitored to identify if any additional opioids prescriptions were provided by any provider

SECONDARY OUTCOMES:
Post-operative pain after discharge | 7 days
  Visual analog pain scale (which ranges from 0-10) will be completed daily for 7 days. Score of zero signifies no pain at all and a a score of 10 implies the worst pain ever experienced.
Satisfaction score during home recovery | 7 days
  Overall satisfaction score (0-100%) with post-operative pain, discomfort and recovery at home. A higher score signifies more satisfaction with pain control during the recovery process.
Contact with healthcare facilities | 30 days
  All phone calls to the clinic, unplanned visits, emergency room visits, hospital admissions will recorded and combined as a single measure of contact with any healthcare facility as a measure of resource utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Badar Mian, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No